CLINICAL TRIAL: NCT06118047
Title: Efficacy and Safety of Crisaborole Ointment, a Phosphodiesterase 4 (PDE4) Inhibitor, for the Topical Treatment of Cetuximab-Related Skin Toxicity Among Metastatic Colorectal Cancer Patients：A Prospective, Single-arm, Phase II Clinical Trial
Brief Title: Crisaborole Ointment for Skin Toxicity Induced by Cetuximab
Acronym: COSTIC
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, WeiWei Xiao, Chief physician, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: B2022-648
Record Dates: First submitted 2023-10-31; First posted 2023-11-07 (Actual); Last update posted 2023-11-07 (Actual); Status verified 2023-07

CONDITIONS: Metastatic Colorectal Cancer; Cetuximab; Skin Toxicity
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Cetuximab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention group (Experimental): crisaborole ointment
  Interventions: Drug: Crisaborole Ointment; Drug: Cetuximab

INTERVENTIONS:
Drug: Crisaborole Ointment — Crisaborole ointment to be applied twice daily.
Drug: Cetuximab — Cetuximab

SUMMARY:
This is a prospective, single-arm, phase II clinical trial that will enroll metastatic colorectal cancer patients with Cetuximab-Related Skin Toxicity, who will receive crisaborole ointment twice daily.

DETAILED DESCRIPTION:
The efficacy of cetuximab has been demonstrated in treating metastatic colorectal cancer (mCRC). Skin toxicities, especially acneiform eruption, are the major side effects associated with cetuximab, which affect patients' quality of life and can lead to treatment discontinuation and cetuximab dose reduction.

This prospective, single-arm, phase II clinical trial aims to explore the efficacy and safety of crisaborole ointment in Cetuximab-Related Skin Toxicity. A total of 33 mCRC patients with acneiform eruption will be enrolled. All of the participants will receive crisaborole ointment twice daily. The total follow-up time is 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosed mCRC and undergoing Cetuximab treatment;
2. ≥2 grade EGFR inhibitor-related acneiform eruption, evaluated by National Cancer Institute (NCI) Common Terminology Criteria Adverse Events (CTCAE）5.0;
3. Age 18 years and older；
4. ECOG performance status 0-2.；
5. Bone marrow ,brain, heart, kidney and other organ function well;；
6. Expected survival time more than 3 months;

Exclusion Criteria:

1. The presence of any active skin disease；
2. Undergoing any current hormone therapy for any other disease;
3. Prior allergic reaction or severe intolerance to crisaborole ointment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Estimated)
Dates: Start 2023-08-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Remission rate of EGFR inhibitor-related acneiform eruption | From date of randomization until the date of remission，assessed up to 8 weeks.
  Grading of acneiform eruption would be assessed according to National Cancer Institute (NCI) Common Terminology Criteria Adverse Events (CTCAE) 5.0. Remission was defined as a reduction in acneiform eruption from grade 2 to grade 1 or grade 3 to grade 2 sustained for at least 2 weeks.

SECONDARY OUTCOMES:
Remission time of EGFR inhibitor-related acneiform eruption | From date of randomization until the date of remission，assessed up to 8 weeks.
  Grading of acneiform eruption would be assessed according to NCI-CTCAE 5.0. Remission was defined as a reduction in acneiform eruption from grade 2 to grade 1 or grade 3 to grade 2 sustained for at least 2 weeks
Cetuximab treatment discontinuation rate | 8 weeks from randomization.
  Rate of Cetuximab treatment discontinuation due to skin toxicity
Cetuximab dose reduction rate | 8 weeks from randomization.
  Rate of Cetuximab dose reduction due to skin toxicity
Level of paronychia, xeroderma and pruritus | 8 weeks from randomization.
  Grading of paronychia, xeroderma and pruritus would be assessed according to NCI-CTCAE 5.0.
Quality of life (FACT-EGFRI-18) | The 0,2,4,6,8,10,12 weeks from randomization.
  Functional Assessment of Cancer Therapy （FACT）questionnaire to assess dermatologic symptoms associated with epidermal growth factor receptor inhibitors （FACT-EGFRI-18）
Quality of life（EORTC QLQ-C30) | The 0,2,4,6,8,10,12 weeks from randomization.
  Questionnaire of the European Organisation for Research and Treatment of Cancer quality of life (EORTC QLQ-C30)

CONTACTS AND LOCATIONS:
Overall Officials: Weiwei Xiao, Principal Investigator — Sun Yat-sen University
Locations (1):
- WeiWei Xiao, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Kim YS, Ji JH, Oh SY, Lee S, Huh SJ, Lee JH, Song KH, Son CH, Roh MS, Lee GW, Lee J, Kim ST, Kim CK, Jang JS, Hwang IG, Ahn HK, Park LC, Oh SY, Kim SG, Lee SC, Lim DH, Lee SI, Kang JH. A Randomized Controlled Trial of Epidermal Growth Factor Ointment for Treating Epidermal Growth Factor Receptor Inhibitor-Induced Skin Toxicities. Oncologist. 2020 Jan;25(1):e186-e193. doi: 10.1634/theoncologist.2019-0221. Epub 2019 Sep 6. PMID 31492766
- [Background] Klufa J, Bauer T, Hanson B, Herbold C, Starkl P, Lichtenberger B, Srutkova D, Schulz D, Vujic I, Mohr T, Rappersberger K, Bodenmiller B, Kozakova H, Knapp S, Loy A, Sibilia M. Hair eruption initiates and commensal skin microbiota aggravate adverse events of anti-EGFR therapy. Sci Transl Med. 2019 Dec 11;11(522):eaax2693. doi: 10.1126/scitranslmed.aax2693. PMID 31826981
- [Background] Hofheinz RD, Lorenzen S, Trojan J, Ocvirk J, Ettrich TJ, Al-Batran SE, Schulz H, Homann N, Feustel HP, Schatz M, Kripp M, Schulte N, Tetyusheva M, Heeger S, Vlassak S, Merx K. EVITA-a double-blind, vehicle-controlled, randomized phase II trial of vitamin K1 cream as prophylaxis for cetuximab-induced skin toxicity. Ann Oncol. 2018 Apr 1;29(4):1010-1015. doi: 10.1093/annonc/mdy015. PMID 29360920
- [Background] Pinto C, Barone CA, Girolomoni G, Russi EG, Merlano MC, Ferrari D, Maiello E; American Society of Clinical Oncology; European Society of Medical Oncology. Management of skin toxicity associated with cetuximab treatment in combination with chemotherapy or radiotherapy. Oncologist. 2011;16(2):228-38. doi: 10.1634/theoncologist.2010-0298. Epub 2011 Jan 27. PMID 21273511
- [Background] Pinto C, Barone CA, Girolomoni G, Russi EG, Merlano MC, Ferrari D, Maiello E. Management of Skin Reactions During Cetuximab Treatment in Association With Chemotherapy or Radiotherapy: Update of the Italian Expert Recommendations. Am J Clin Oncol. 2016 Aug;39(4):407-15. doi: 10.1097/COC.0000000000000291. PMID 27077276